CLINICAL TRIAL: NCT04110652
Title: Effect of a Pulmonary Rehabilitation Program on Hospital Mortality and Disability in Patients With Acute Ischemic Stroke
Brief Title: Effect of Pulmonary Rehabilitation Program on Patients With Acute Ischemic Stroke, Mortality and Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Collaborators: Mohamed Wahid Elsayed Elsayed (Unknown); Prof. Dr. Tamer Abdullah Helmy (Unknown); Dr. Osama Saeed Hassan (Unknown)
Responsible Party: Principal Investigator, Rehab Abdelaal ELnemr, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0105838
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Stroke, Acute; Pulmonary Rehabilitation; Morality
Keywords: stroke; rehabilitation; mortality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Active Comparator): 40 patients with acute stroke will receive Stroke management based on the guidelines of the American Heart Association/American Stroke Association.(20-22) in addition to pulmonary rehabilitation program.
  Interventions: Other: pulmonary rehabilitation program
- control group (Placebo Comparator): 40 patients with acute stroke will receive Stroke management based on the guidelines of the American Heart Association/American Stroke Association.
  Interventions: Other: pulmonary rehabilitation program

INTERVENTIONS:
Other: pulmonary rehabilitation program — The pulmonary rehabilitation program consisting of inspiratory muscle training, manual hyperinflation. chest wall mobilization, rib-cage compression, cough function training, postural drainage and secretion removal will be applied to patient group.
  The program will be conducted by physical therapists for 30-45 minutes daily during ICU stay.
  The exercise intensity will be increased gradually over the course. Each patient's performance during the exercise sessions will be recorded and reported regularly.

SUMMARY:
Severe stroke remains an important cause of mortality and morbidity, despite advances in disease management, acute treatment and secondary measures. Among all post-stroke complications, pneumonia constitutes a major complication with a strong impact on morbidity and mortality. Research also showed that a reduction in respiratory muscle and abdominal muscle strength contributed to pulmonary and respiratory dysfunction following a stroke. Low respiratory muscle function decreases the efficacy of rehabilitation because it leads to exercise intolerance in stroke patients. Thus, special exercise programs are needed to improve the pulmonary function and respiratory muscle strength of stroke patients The aim of pulmonary rehabilitation program is to enhance respiratory muscle resistance during breathing, thereby improving respiratory function. Previous studies demonstrated that pulmonary rehabilitation programs improved respiratory functions in cardiac disease and chronic obstructive pulmonary disease patients

DETAILED DESCRIPTION:
The study will be conducted on 80 adult patients with Acute Ischemic Stroke.

Inclusion criteria:

* Adult (≥18 years old).
* With Acute Ischemic Stroke.

Exclusion criteria:

* Hemorrhagic stroke.
* GCS < 7 on admission.
* Clinical signs of infection on admission.
* Significant pulmonary disease, angina, myocardial infarction or acute heart failure within three months.

For every eligible patient the following data will be collected:

* Demographic data including age & sex.
* Vital signs.
* Glasgow Coma Score on admission after primary respiratory and hemodynamic stabilization.
* Stroke severity on admission assessed by the National Institute of Health Stroke Scale (NIHSS).
* All patients will undergo a CT scan of the brain on admission. Diagnostic procedures such as Doppler ultrasound of the carotid arteries, MRI, and echocardiography will be ordered if deemed necessary by the treating physician.
* Stroke subtype classification utilizing both the TOAST (Trial of ORG 10172 in Acute Stroke Treatment) method and The Oxfordshire Community Stroke Project.
* Pre-existing comorbid conditions (any treatment and/or patient's self-report): Hypertension, Diabetes Mellitus, Atrial Fibrillation, COPD, CHF, and Current Smoking.
* Evidence for any type of dysphagia documented by a standardized dysphagia screening test.
* Laboratory data: White Blood Cell (WBC) Count, C-reactive Protein (CRP), and Blood Glucose will be done daily.

Grouping The patients will be randomized into 2 groups by conventional method of randomization where patients in group 1 (control group) will be selected in odd numbers and those in group 2 (patients receiving pulmonary rehabilitation program) will be selected in even numbers.

Stroke management Group 1: (Control group) 40 patients will receive Stroke management based on the guidelines of the American Heart Association/American Stroke Association.

Group 2: (Patients receiving pulmonary rehabilitation program) 40 patients will receive Stroke management based on the guidelines of the American Heart Association/American Stroke Association in addition to pulmonary rehabilitation program.

Enrolled patients will be prospectively followed up for:

1. Primary outcome:

   • The diagnosis of pneumonia within the first 7 days after admission. (Diagnosis will be made according to modified criteria of the CDC
2. Secondary outcome:

   * In-hospital or 30 days mortality.
   * Modified Rankin Scale (mRS) at one month.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old).
* With Acute Ischemic Stroke

Exclusion Criteria:

* Hemorrhagic stroke.
* GCS < 7 on admission.
* Clinical signs of infection on admission.
* Significant pulmonary disease, angina, myocardial infarction or acute heart failure within three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-03 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-20 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: The diagnosis of pneumonia within the first 7 days after admission. | within the first 7 days after admission
  Diagnosis will be made according to modified criteria of the CDC

SECONDARY OUTCOMES:
Mortality rate | In-hospital after 30 days
  Modified Rankin Scale (mRS) at one month

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab Abdelaal ELnemr, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
may be after finishing patient collection